## **PATIENT CONSENT FORM**

Study title: Randomised Controlled Trial comparing Metatarsal Method of Transection using Bone Cutters or Bone Saw on Outcomes after Ray Amputation (MetaMet)

| Yes □ | No □ |
|-------|----------------------------------------|
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No□ |
| | Yes |

| FUTURE CONTACT [please choose one or more as you see fit] | | |
|---|---|---|
| <b>OPTION 1:</b> I consent to be re-contacted by researchers about possible | Yes □ | No □ |
| future research <b>related</b> to the current study for which I may be eligible. | | |
| <b>OPTION 2:</b> I consent to be re-contacted by researchers about possible | | No □ |
| future research <b>unrelated</b> to the current study for which I may be eligible. | | |

## To be completed by the trial participant.

| | | I | l |
|---|---|---|---|
| Patient Name (Block Capit | als) | Patient Signature | Date |
| Translator Name (Block Ca | <br>pitals) | <br>Translator Signature | <br>Date |
| Legal Representative/Guardian Name | | Legal Representative/Gu | ardian Signature Date |
| purpose of this study in a | aken the time<br>way that they | tigator or nominee. to fully explain to the above could understand. I have exp ed them to ask questions on | lained the risks involved as |
| Name (Block Capitals) | <br><br> Qualifica | <br>tions Signature | <br><br> Date |
| Name (Block Capitals) 3 copies to be made: 1 for | · | tions Signature PI and 1 for hospital records | Date |